CLINICAL TRIAL: NCT05125315
Title: Intraoperative Hemodynamics in Patients Undergoing Coronary Artery Bypass Graft for Long-term Outcom
Brief Title: Intraoperative Hemodynamics in CABG
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, Jun Ma, Directer of anesthesia department, Beijing Anzhen Hospital
Other Study IDs: 2021-1101
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- low-hemosynamics
- high-hemodynamics

SUMMARY:
The study is to determine the effects of the intraoperative hemodynamics in patients undergoing coronary artery bypass graft on the short-term and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* age18-80 for CABG surgery only

Exclusion Criteria:

* Emergency surgery atrial fibrillation using ECMO/VAD

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing isolated CABG will included in this study. All the ertracted patients are ethnic Chinese. Patients undergoing emergency surgery or using ECOM/VAD will be excluded.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
long-time motality after CABG | 1 year
  To determine the motality in patients undergoing CABG after 1 year